CLINICAL TRIAL: NCT03945526
Title: Effect of Astaxanthin Supplementation on Plasma Malondialdehyde Levels and National Institute of Health Stroke Scale Score of Acute Ischemic Stroke Patients: A Randomized Trial
Brief Title: Effect of Astaxanthin Supplementation on Plasma Malondialdehyde Levels and NIHSS of Stroke Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Gabriella Nurahmani Putri, Assistant Clinical Nutrition Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neuronutrition
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Cerebral Stroke; Malondialdehyde; Oxidative Stress
Keywords: Astaxanthin; Antioxidant; Plasma Malondialdehyde; NIHSS score; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — astaxanthine

STUDY DESIGN:
Intervention Model Description: Astaxanthin and Placebo
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin (Active Comparator): Astaxanthin supplementation will be given at 2 x 8mg for 7 days.
  Interventions: Drug: Astaxanthine
- Control (Placebo Comparator): A placebo will be given, which takes the form of a drug with the exact same shape and color as astaxanthin supplementation
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Astaxanthine
  Other Names: Astaxanthine 8mg
  Arms: Astaxanthin
Drug: Placebo Oral Tablet
  Other Names: Astaxanthine placebo
  Arms: Control

SUMMARY:
This is an interventional randomized, controlled trial in analyzing the effects of astaxanthin supplementation on plasma malondialdehyde levels and NIHSS of acute ischemic stroke patients. According to published studies, it was hypothesized that acute ischemic stroke patients who were given astaxanthin would have lower plasma malondialdehyde levels and lower NIHSS score compared to the control group.

DETAILED DESCRIPTION:
There were a total of 24 subjects, with 12 subjects in the intervention group and 12 subjects in the control group.The participants were divided into an interventional group and a control group. The interventional group was given astaxanthin supplementation 2 x 8mg per day for 7 days, while the control group was given placebo.

ELIGIBILITY:
Inclusion Criteria:

* 40-65 years old
* Has acute ischemic stroke with an onset of less than 48 hours before hospital admission
* NIHSS score of less than or equal to 15
* Can consume food orally or enterally
* Has given their consent to be a participant in the study

Exclusion Criteria:

* Renal failure
* Liver failure
* Is taking supplements other than his or her main stroke medications
* Has taken antioxidant supplements in the last 3 months before stroke onset

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03-23 (Actual); Primary Completion 2010-06-09 (Actual); Study Completion 2010-06-09 (Actual)

PRIMARY OUTCOMES:
Plasma Malondialdehyde Levels on Astaxanthine Treated Stroke Patients as Assessed by Wills Spectrophotometry | 7 days
  This method used Thiobarbituric acid reaction (TBAR) with substances such as malondialdehyde. The scale was 0.367 nmol/ml-0.707 nmol/ml. The value above 0.707nmol/ml would be the worse outcome, and value less than 0.367nmol/ml would be the best outcome. Bivariate analysis was used to analyze the results (T-test or the Mann-Whitney Test).
National Institute of Health Stroke Scale on Astaxanthine Treated Stroke Patients | 7 days
  Score scale was 4-15, where less than 4 indicates mild neurologic deficit, 4-15 moderate neurologic deficit, and more than 15 severe neurologic deficit. They will be assessed before and after the trial to compare how each participant improved after given the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Salim Harris, SpS, Study Chair — IDI; Sri Sukmaniah, SpGK, Study Chair — IDI
Locations (1):
- Department of Nutrition University of Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber PA, Demchuk AM, Hirt L, Buchan AM. Biochemistry of ischemic stroke. Adv Neurol. 2003;92:151-64. No abstract available. PMID 12760178
- [Background] Shen H, Kuo CC, Chou J, Delvolve A, Jackson SN, Post J, Woods AS, Hoffer BJ, Wang Y, Harvey BK. Astaxanthin reduces ischemic brain injury in adult rats. FASEB J. 2009 Jun;23(6):1958-68. doi: 10.1096/fj.08-123281. Epub 2009 Feb 13. PMID 19218497
- [Background] Palozza P, Krinsky NI. Astaxanthin and canthaxanthin are potent antioxidants in a membrane model. Arch Biochem Biophys. 1992 Sep;297(2):291-5. doi: 10.1016/0003-9861(92)90675-m. PMID 1497349
- [Background] Hussein G, Nakamura M, Zhao Q, Iguchi T, Goto H, Sankawa U, Watanabe H. Antihypertensive and neuroprotective effects of astaxanthin in experimental animals. Biol Pharm Bull. 2005 Jan;28(1):47-52. doi: 10.1248/bpb.28.47. PMID 15635162
- [Background] Gariballa SE, Sinclair AJ. Assessment and treatment of nutritional status in stroke patients. Postgrad Med J. 1998 Jul;74(873):395-9. doi: 10.1136/pgmj.74.873.395. PMID 9799909
- [Background] Demirkaya S, Topcuoglu MA, Aydin A, Ulas UH, Isimer AI, Vural O. Malondialdehyde, glutathione peroxidase and superoxide dismutase in peripheral blood erythrocytes of patients with acute cerebral ischemia. Eur J Neurol. 2001 Jan;8(1):43-51. doi: 10.1046/j.1468-1331.2001.00166.x. PMID 11509080